CLINICAL TRIAL: NCT04850781
Title: Home-delivered Meals for Persons With Dementia: Which Model Delays Nursing Home Placement?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Meals on Wheels America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2008002788; R61AG070170 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-20 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Dementia
Keywords: Nutrition; Homebound; Food insecurity
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a Phase 1 pilot feasibility study that uses an embedded, pragmatic randomized clinical trial design.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Meals (Active Comparator): A lunch-time meal delivered to participants' homes multiple times per week with wellness check and socialization.
  Interventions: Behavioral: Daily home meal delivery
- Frozen, Drop-shipped Meals (Experimental): 10 frozen meals that are mailed to participants every two weeks.
  Interventions: Behavioral: Bi-weekly frozen meal home delivery

INTERVENTIONS:
Behavioral: Bi-weekly frozen meal home delivery — All participants randomized to this arm will receive 10 frozen meals that are mailed to their home every two weeks from a MOW vendor, TRIO foods.
  Arms: Frozen, Drop-shipped Meals
Behavioral: Daily home meal delivery — All participants randomized to this arm will receive meals delivered to their home multiple times per week from a MOW program employee/volunteer with a wellness check and socialization.
  Arms: Daily Meals

SUMMARY:
This project is the pilot phase of a pragmatic randomized clinical trial comparing outcomes among older adults with Alzheimer's disease and related dementias (ADRD) receiving home-delivered meals. This pilot will test and validate vital elements and procedures including: 1) enrolling persons with ADRD on Meals on Wheels (MOW) programs' waiting lists to receive one of the two types of meals; 2) recruiting a subsample of participants and caregivers to participate in telephone interviews; 3) extracting and transferring program data to Brown University; 4) linking participant data with Medicare and nursing home assessment data. Persons with ADRD receiving meals and their caregivers will be recruited to pilot interview guides. The interviews will provide important process and mechanistic information about the experiences receiving meals and participants' outcomes.

DETAILED DESCRIPTION:
236 individuals on the waiting list at three MOW programs (Neighborly Senior Services in Clearwater, Florida; Visiting Nurse Association of Texas in Dallas, Texas; Meals on Wheels - San Antonio in San Antonio, Texas) will be randomized to one of the following modes of delivery: 1) meals that are delivered multiple times per week by a MOW program volunteer or paid driver and includes socialization and a wellness check or 2) frozen meals that are mailed to participants' homes every two weeks. Persons with ADRD receiving meals and their caregivers will be recruited to pilot interview guides.

The primary aim is to test and validate procedures to recruit participants with ADRD and evaluate their outcomes in partnership with MOW programs. The study also aims to characterize differences in the processes and potential mechanisms contributing to outcomes between the two modes of meal delivery among older adults with ADRD. The qualitative interviews with participants and their caregivers will provide important process and mechanistic information about the experiences receiving meals and participants' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* On MOW program waiting list
* 66 years of age or older (to allow for Medicare enrollment and a one-year baseline look-back)
* Self-reporting a diagnosis of memory loss, dementia, cognitive impairment, or Alzheimer's disease

Exclusion Criteria:

* Residing in a service area where it is not possible to receive the daily-delivered meals.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 243 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kali S Thomas, PhD, Principal Investigator — Brown University, School of Public Health
Locations (3):
- United States (3):
  - Neighborly Senior Services, Clearwater, Florida
  - Visiting Nurse Association of Texas, Dallas, Texas
  - Meals on Wheels - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bunker JN, Hilgeman MM, McCreedy E, Gadbois E, Thomas KS. Evaluating the Implementation Fidelity of a Pilot Pragmatic Randomized Clinical Trial Comparing Daily-Delivered Meals to Mailed Frozen Meals. J Appl Gerontol. 2024 Nov;43(11):1605-1610. doi: 10.1177/07334648241248269. Epub 2024 Apr 30. PMID 38686741
- [Derived] Thomas KS, Bunker J, Gadbois E, Hilgeman M, McCreedy E, Mills W, Ornstein KA, Reckrey J, Gutman R. Home-Delivered Meals and Nursing Home Placement Among People With Self-Reported Dementia: A Pilot Pragmatic Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2347195. doi: 10.1001/jamanetworkopen.2023.47195. PMID 38117500
- [Derived] Gadbois EA, Bunker JN, Hilgeman M, Shield R, McAuliff KE, Mills W, Thomas K. Feasibility of conducting qualitative research with persons living with dementia and their caregivers during a home-delivered meals pilot trial. Pilot Feasibility Stud. 2023 Apr 22;9(1):65. doi: 10.1186/s40814-023-01302-5. PMID 37085899
- See also: Peer-reviewed paper describing the results from the qualitative sub-study — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-023-01302-5

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants at 3 home-delivered meals sites were identified based on 1) being on a waitlist 2) self-identifying as having dementia and 3) being age 66 years and older. Randomization and enrollment began in April 2021 and continued until September 2021
Pre-assignment Details: 243 participants were enrolled in the trial.
Period: Overall Study
Arm/Group | Daily Meals | Frozen, Drop-shipped Meals
Started | 128 | 115
Completed | 128 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was an intent-to-treat design; meaning, all participants who were enrolled were analyzed, regardless of how long they received meals.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Meals | Frozen, Drop-shipped Meals | Total
Number analyzed (Participants) | 128 | 115 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 128 | 115 | 243
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 78 | 152
  Male | 54 | 37 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 21 | 22 | 43
  White | 64 | 64 | 128
  Hispanic | 37 | 25 | 62
  Other | 6 | 4 | 10
Lives Alone [Count of Participants; unit: Participants] | 53 | 66 | 119

OUTCOME MEASURES:

1. Primary Outcome: Time to Nursing Home Placement
Description: We report the restricted mean survival time, which is the average time free from an event (i.e., nursing home placement) up until 180 days or death, whichever comes first.
Time Frame: 6 months / 180 days
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Daily Meals | Frozen, Drop-shipped Meals
Number analyzed (Participants) | 128 | 115
Days | 172.0725 [168.8933 to 175.2517] | 165.0270 [161.1035 to 168.9505]

ADVERSE EVENTS:
Time Frame: 6 months from randomization/
Description: All-cause Mortality - sites reported deaths
  SAE - no SAEs were expected, as intervention does not contain any components with the potential to be life threatening, require or prolong hospitalization, cause persistent or significant disability or incapacity, or result in congenital anomalies or birth defects.
  AEs - the potential AEs that could occur during this trial are mild distress, negative emotional reactions, or confusion in response to being interviewed by a data collector.
Arm/Group | Daily Meals | Frozen, Drop-shipped Meals
All-Cause Mortality (participants affected / at risk) | 5/128 | 8/115
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/115
Other Adverse Events (participants affected / at risk) | 0/128 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-11-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT04850781/Prot_SAP_ICF_001.pdf